CLINICAL TRIAL: NCT04353544
Title: Effect of Delayed vs Immediate Umbilical Cord Clamping on Maternal Blood Loss in Term Spontaneous Vaginal Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: Casa di Cura Accreditata Fabia Mater, Rome, Italy (Unknown)
Responsible Party: Principal Investigator, Gabriele Saccone, principal investigator, medical doctor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1/04-18OST
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate cord clamping (Active Comparator): Immediate cord clamping was defined as clampingwithin 15 seconds of birth
  Interventions: Other: delayed cord clamping
- delayed cord clamping (Experimental): when the cord stopped pulsing, or five minutes
  Interventions: Other: delayed cord clamping

INTERVENTIONS:
Other: delayed cord clamping — delayed cord clamping

SUMMARY:
Policies for timing of cord clamping vary, with early cord clamping generally carried out in the first 60 seconds aLer birth, whereas latercord clamping usually involves clamping the umbilical cord greater than one minute after the birth or when cord pulsation has ceased

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* at term
* cephalic presentation
* spontaneous labor
* spontaneous vaginal delivery

Exclusion Criteria:

* multiple gestation
* preterm gestation
* induced labor
* operative delivery
* hypertension or preeclampsia
* fetal anomaly
* abnormal placentation
* planned cord blood banking
* maternal bleeding disorder

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 122 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
change in maternal hemoglobin level on post delivery day 1 compared with the predelivery hemoglobin level | day 1 after delivery
  The primary outcome was an objective measure of maternal blood loss: the change in maternal hemoglobin level on postdelivery day 1 compared with the predelivery hemoglobin level.

SECONDARY OUTCOMES:
postpartum hemorrhage | at the time of delivery
  defined as estimated blood loss>500cc
uterotonic administration | at the time of delivery
need for blood transfusion | at the time of delivery
jaundice | day 10 of life
  neonatal jaundice

CONTACTS AND LOCATIONS:
Locations (1):
- Casa di Cura Accreditata Fabia Mater, Rome, Italy, Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided
not planned

REFERENCES:
- [Derived] De Angelis C, Saccone G, Sorichetti E, Alagna M, Zizolfi B, Gragnano E, Legnante A, Sardo ADS. Effect of delayed versus immediate umbilical cord clamping in vaginal delivery at term: A randomized clinical trial. Int J Gynaecol Obstet. 2022 Dec;159(3):898-902. doi: 10.1002/ijgo.14223. Epub 2022 May 2. PMID 35428979